CLINICAL TRIAL: NCT03759041
Title: ECO-RESET: A Phase 2B, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose, Multicenter Study to Assess Efficacy and Safety of SER-287 in Adults With Active Mild-to-Moderate Ulcerative Colitis
Brief Title: A Study to Assess Efficacy and Safety of SER-287 in Adults With Active Mild-to-Moderate Ulcerative Colitis
Acronym: ECO-RESET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the lack of a clinical efficacy signal in the induction treatment phase, Seres closed the dosing phases of open label and maintenance portions of the study. Patients who had received prior doses were followed for safety data.
Sponsor: Seres Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SERES-201
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-07

CONDITIONS: Ulcerative Colitis
Keywords: microbiome
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (after placebo pre-treatment) (Placebo Comparator): Once-daily dosing of Placebo (after placebo pre-treatment)
  Interventions: Drug: Placebo for Vancomycin Pre-Treatment; Drug: Placebo for SER-287
- SER-287 Induction Dosing (after vancomycin pre-treatment) (Experimental): Once-daily dosing of SER-287 (Induction Dose, after vancomycin pre-treatment)
  Interventions: Drug: Vancomycin Pre-Treatment; Drug: SER-287
- SER-287 Step-Down Induction Dosing (after vancomycin pre-treatment) (Experimental): Once-daily dosing of SER-287 (Step-Down Induction Dose, after vancomycin pre-treatment)
  Interventions: Drug: Vancomycin Pre-Treatment; Drug: SER-287

INTERVENTIONS:
Drug: Vancomycin Pre-Treatment — Four times per day dosing of vancomycin pre-treatment
  Arms: SER-287 Induction Dosing (after vancomycin pre-treatment); SER-287 Step-Down Induction Dosing (after vancomycin pre-treatment)
Drug: Placebo for Vancomycin Pre-Treatment — Four times per day dosing of placebo pre-treatment
  Arms: Placebo (after placebo pre-treatment)
Drug: SER-287 — Once-daily dosing of SER-287
  Other Names: Eubacterial Spores, Purified Suspension, Encapsulated
  Arms: SER-287 Induction Dosing (after vancomycin pre-treatment); SER-287 Step-Down Induction Dosing (after vancomycin pre-treatment)
Drug: Placebo for SER-287 — Once-daily dosing of Placebo for SER-287
  Arms: Placebo (after placebo pre-treatment)

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose, Multicenter Study to Assess Efficacy and Safety of SER-287 in Adults with Active Mild-to-Moderate Ulcerative Colitis

DETAILED DESCRIPTION:
This is a Phase 2B randomized, double-blind, placebo-controlled, multiple dose, multicenter study designed to evaluate the efficacy, safety and microbiome alterations associated with two dose levels of SER-287, after pre-treatment with vancomycin, in adult subjects, age 18-80, with active mild-to-moderate ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of UC at least three months prior to screening, and with a minimum disease extent of 15 cm from the anal verge
* Active mild-to-moderate UC
* Inadequate response to, loss of response to, or intolerance of, at least one of the following conventional therapies: 5-ASA compounds, corticosteroids, 6-mercaptopurine (6-MP) or azathioprine (AZA), anti-TNFα, anti-integrin or tofacitinib

Exclusion Criteria:

* Known history of Crohn's disease
* No previous history of treatment for UC (treatment-naïve)
* Subjects on steroid medication who are unable to have steroids tapered and be completely off steroids at least two weeks prior to screening
* Unable to stop steroid enemas or suppositories, or 5-ASA enemas or suppositories, at least two weeks prior to screening
* Subjects who have received any investigational or approved biologic therapy within eight weeks or five half-lives prior to screening (whichever is longer)
* Subjects who have received any investigational or approved non-biologic therapy, except for those specifically listed in the Permitted Concomitant Medications, for the treatment of underlying disease, within 30 days or five half-lives prior to screening (whichever is longer)
* Major gastrointestinal surgery (not including appendectomy or cholecystectomy) within two months before screening, or any history of total colectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa von Moltke, MD, Study Director — Seres Therapeutics, Inc.
Locations (83):
- United States (73):
  - (Investigator site), Phoenix, Arizona
  - (Investigator site), North Little Rock, Arkansas
  - (Investigator site), La Jolla, California
  - (Investigator site), Lancaster, California
  - (Investigator site), Los Angeles, California
  - (Investigator site), Mountain View, California
  - (Investigator site), San Diego, California
  - (Investigator site), Wheat Ridge, Colorado
  - (Investigator site), Danbury, Connecticut
  - (Investigator site), Hamden, Connecticut
  - (Investigator site), Boca Raton, Florida
  - (Investigator site), Clearwater, Florida
  - (Investigator site), Crystal River, Florida
  - (Investigator site), Fort Lauderdale, Florida
  - (Investigator site), Hialeah, Florida
  - (Investigator site), Jacksonville, Florida
  - (Investigator site), Miami, Florida
  - (Investigator site), Naples, Florida
  - (Investigator site), Ocala, Florida
  - (Investigator site), Orlando, Florida
  - (Investigator site), Pompano Beach, Florida
  - (Investigator site), Port Orange, Florida
  - (Investigator site), Tampa, Florida
  - (Investigator site), Athens, Georgia
  - (Investigator site), Atlanta, Georgia
  - (Investigator site), Marietta, Georgia
  - (Investigator site), Chicago, Illinois
  - (Investigator site), Indianapolis, Indiana
  - (Investigator site), Lexington, Kentucky
  - (Investigator site), Lake Charles, Louisiana
  - (Investigator site), Metairie, Louisiana
  - (Investigator site), Monroe, Louisiana
  - (Investigator site), New Orleans, Louisiana
  - (Investigator site), Shreveport, Louisiana
  - (Investigator site), Baltimore, Maryland
  - (Investigator site), Glen Burnie, Maryland
  - (Investigator site), Ann Arbor, Michigan
  - (Investigator site), Farmington Hills, Michigan
  - (Investigator site), Rochester, Minnesota
  - (Investigator site), Bridgeton, Missouri
  - (Investigator site), Creve Coeur, Missouri
  - (Investigator site), Las Vegas, Nevada
  - (Investigator site), Reno, Nevada
  - (Investigator site), Lebanon, New Hampshire
  - (Investigator site), Great Neck, New York
  - (Investigator site), Hartsdale, New York
  - (Investigator site), New York, New York
  - (Investigator site), Asheville, North Carolina
  - (Investigator site), Chapel Hill, North Carolina
  - (Investigator site), Durham, North Carolina
  - (Investigator site), Raleigh, North Carolina
  - (Investigator site), Winston-Salem, North Carolina
  - (Investigator site), Cincinnati, Ohio
  - (Investigator site), Oklahoma City, Oklahoma
  - (Investigator site), Columbia, South Carolina
  - (Investigator site), Greenville, South Carolina
  - (Investigator site), Memphis, Tennessee
  - (Investigator site), Nashville, Tennessee
  - (Investigator site), Bedford, Texas
  - (Investigator site), Fort Sam Houston, Texas
  - (Investigator site), Houston, Texas
  - (Investigator site), McAllen, Texas
  - (Investigator site), San Antonio, Texas
  - (Investigator site), Temple, Texas
  - (Investigator site), Ogden, Utah
  - (Investigator site), Salt Lake City, Utah
  - (Investigator site), Leesburg, Virginia
  - (Investigator site), Lynchburg, Virginia
  - (Investigator site), Reston, Virginia
  - (Investigator site), Richmond, Virginia
  - (Investigator site), Spokane, Washington
  - (Investigator site), Madison, Wisconsin
  - (Investigator site), Milwaukee, Wisconsin
- Canada (10):
  - (Investigator site), Edmonton, Alberta
  - (Investigator site), New Westminster, British Columbia
  - (Investigator site), Bridgewater, Ontario
  - (Investigator site), Greater Sudbury, Ontario
  - (Investigator site), Lindsay, Ontario
  - (Investigator site), London, Ontario
  - (Investigator site), Toronto, Ontario
  - (Investigator site), Vaughan, Ontario
  - (Investigator site), Greenfield Park, Quebec
  - (Investigator site), Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo (After Placebo Pre-treatment) | SER-287 Induction Dosing (After Vancomycin Pre-treatment) | SER-287 Step-Down Induction Dosing (After Vancomycin Pre-treatment)
Started | 69 | 68 | 66
Completed | 42 | 34 | 38
Not Completed | 27 | 34 | 28
Not completed — Withdrawal by Subject | 4 | 10 | 10
Not completed — Adverse Event | 1 | 3 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 15 | 16 | 10
Not completed — Other reason for discontinuation | 0 | 2 | 1
Not completed — Lost to Follow-up | 7 | 2 | 2
Not completed — Subjects did not have a discontinuation page completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (After Placebo Pre-treatment) | SER-287 Induction Dosing (After Vancomycin Pre-treatment) | SER-287 Step-Down Induction Dosing (After Vancomycin Pre-treatment) | Total
Number analyzed (Participants) | 69 | 68 | 66 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (13.24) | 45.7 (14.37) | 44.4 (14.70) | 45.6 (14.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 36 | 34 | 98
  Male | 41 | 32 | 32 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 6 | 23
  Not Hispanic or Latino | 61 | 57 | 59 | 177
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 6 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 3 | 6 | 18
  White | 56 | 59 | 55 | 170
  More than one race | NA — Data not collected | NA — Data not collected | NA — Data not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 12 | 7 | 27
  United States | 61 | 56 | 59 | 176

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission (Count of Participants)
Description: Clinical remission for the induction treatment period:
  * Stool Frequency subscore = 0 or 1, with at least 1-point decrease from baseline
  * Rectal Bleeding subscore = 0
  * Endoscopic subscore = 0 or 1 on modified Mayo Score, with at least 1-point decrease from baseline
  * No occurrence of UC Flare during the treatment period
  Clinical remission was measured using 3 components of the modified Mayo Score (stool frequency, rectal bleeding and endoscopic subscore), a measure of UC disease activity. These 3 components are each graded from 0 to 3, and are summed together for a composite score, with a higher overall score indicating more severe disease (0 = no disease; 9 = worst disease). The modified Mayo endoscopic subscore excludes friability from an endoscopic subscore of 1.
Time Frame: After 10 weeks of induction dosing
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (After Placebo Pre-treatment) | SER-287 Induction Dosing (After Vancomycin Pre-treatment) | SER-287 Step-Down Induction Dosing (After Vancomycin Pre-treatment)
Number analyzed (Participants) | 69 | 68 | 66
Participants | 8 | 7 | 7

2. Secondary Outcome: Endoscopic Improvement (Count of Participants)
Description: Endoscopic subscore decrease from baseline of at least 1 point, as assessed by flexible sigmoidoscopy or colonoscopy.
  Endoscopic improvement was measured using the modified Mayo Score endoscopic subscore, graded from 0 to 3, with higher scores indicating more severe disease. The modified Mayo endoscopic subscore excludes friability from an endoscopic subscore of 1.
Time Frame: After 10 weeks of induction dosing
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (After Placebo Pre-treatment) | SER-287 Induction Dosing (After Vancomycin Pre-treatment) | SER-287 Step-Down Induction Dosing (After Vancomycin Pre-treatment)
Number analyzed (Participants) | 69 | 68 | 66
Participants | 17 | 17 | 16

ADVERSE EVENTS:
Time Frame: Adverse events presented here are for the 10-week Induction Treatment Period of the study, as well as the 1-week Pre-Treatment Period.
Description: Adverse events are reported for subjects who received any amount of study drug.
Arm/Group | Placebo (After Placebo Pre-treatment) | SER-287 Induction Dosing (After Vancomycin Pre-treatment) | SER-287 Step-Down Induction Dosing (After Vancomycin Pre-treatment)
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/68 | 0/65
Serious Adverse Events (participants affected / at risk) | 1/69 | 3/68 | 1/65
Other Adverse Events (participants affected / at risk) | 6/69 | 23/68 | 12/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (After Placebo Pre-treatment) (N=69) | SER-287 Induction Dosing (After Vancomycin Pre-treatment) (N=68) | SER-287 Step-Down Induction Dosing (After Vancomycin Pre-treatment) (N=65)
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1 | 0
Colon dysplasia (Gastrointestinal disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (After Placebo Pre-treatment) (N=69) | SER-287 Induction Dosing (After Vancomycin Pre-treatment) (N=68) | SER-287 Step-Down Induction Dosing (After Vancomycin Pre-treatment) (N=65)
Colitis ulcerative (Gastrointestinal disorders) | 6 | 8 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 10 | 2
Nausea (Gastrointestinal disorders) | 0 | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Study Protocol (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT03759041/Prot_000.pdf
  • Statistical Analysis Plan: Clinical SAP (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT03759041/SAP_001.pdf
  • Statistical Analysis Plan: Microbiome SAP (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT03759041/SAP_002.pdf